CLINICAL TRIAL: NCT04490213
Title: Scarring At Donor Sites After Split-Thickness Skin Graft: A Prospective, Longitudinal, Randomised Trial; The Observer's View
Brief Title: Scarring At Donor Sites After Split-Thickness Skin Graft.
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Folke Sjoberg, Professor, University Hospital, Linkoeping
Other Study IDs: 2018/212-31
Record Dates: First submitted 2019-09-26; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Donor Site Complication
MeSH Terms: interventions — allevyn; Carboxymethylcellulose Sodium; Motion Pictures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hydrofibre, Aquacel: Study participants were previously treated on their donor sites with these CE-marked dressing products (RCT study published in 2014) and are now compared regarding scar outcome at the donor sites
  Interventions: Other: Allevyn, Aquacel and Tegaderm, Mediskin
- polyurethane foam, Allevyn: Study participants were previolsuy treated on their donor sites with these CE-marked dressing products (RCT study published in 2014) and are now compared regarding scar outcome at the donor sites
  Interventions: Other: Allevyn, Aquacel and Tegaderm, Mediskin
- porcine xenograft, Mediskin: Study participants were previolsuy treated on their donor sites with these CE-marked dressing products (RCT study published in 2014) and are now compared regarding scar outcome at the donor sites
  Interventions: Other: Allevyn, Aquacel and Tegaderm, Mediskin

INTERVENTIONS:
Other: Allevyn, Aquacel and Tegaderm, Mediskin — Wound dressing tested earlier on donor sites, in this study scar outcome between the 3 dressing groups are compared.
  Other Names: polyurethan foam, hydrofibre, film, porcone xenograft

SUMMARY:
The aim of this study was to investigate if previous findings on the association between dressing treatments and subjective opinion on final donor site scar outcome using the patient scale of POSAS could be confirmed objectively.

Scar outcome measurements were assessed by a blinded observer using POSAS and the device: Cutometer dual MPA 580 (Courage and Khazaka Electronic GmbH, Cologne, Germany) to measure the viscoelasticity of the skin.

DETAILED DESCRIPTION:
This is the third and last part of a clinical project concerning the treatment of split thickness skin graft donor sites. In the first part the Investigators completed a randomised clinical trial (RCT) in which donor sites were randomly assigned to treatment with either hydrofibre covered with film, non-adhesive polyurethane foam, or porcine xenograft. Results from the first study indicated that donor sites treated with hydrofibre and porcine xenograft healed significantly faster than those treated with polyurethane foam. As the hydrofibre was the most comfortable, easy to use, and cost-effective it was implemented as the standard of care for donor sites at the specific centre.

In the initial RCT, patients treated with polyurethane foam showed significantly longer healing times than the other treatment groups. As longer healing time has been shown to be a predictor for pathological donor site scarring it was hypothesised that this group would be the most unsatisfied with their scars, if they had any donor site scar at all eight years after their skin graft. In the second part of the project the long-term scar outcomes of the donor sites included in the RCT was investigated. Study participants were asked to evaluate their scars using the "Patients part" of the Patient and Observer Scar Scale (POSAS). After analysing the data collected in the second part, it was concluded that the fast and moist healing seen with hydrofibre seemed to result in significantly more satisfied patients - and members of the polyurethane foam group, as hypothesised, were significantly more unsatisfied with their donor site scars. The Investigators also found that the dressing associated with the fastest wound healing (the porcine xenograft) also had the poorest long-term outcome for scarring, according to the patients' opinion. This contradicts what is claimed to be the relation between duration of healing and donor site scarring.

In this last, third study, the aim was to investigate if the previous findings could be confirmed by an evaluation done by a blinded observer using POSAS. Donor sites were also evaluated for firmness and elasticity using the device; Cutometer dual MPA 580 (Courage and Khazaka Electronic GmbH, Cologne, Germany), which is described in the Method section.

ELIGIBILITY:
Inclusion Criteria:

Participation in part I (RCT) and part II of the project

Exclusion Criteria:

No former participation in the project

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Of the 27 participants in the second part of the study, two had died, six (with a total of 8 donor sites) chose not to participate and two did not answer our letter. The remaining 17 were included in the Observer follow up. Of the 17 participants, five came from the hydrofibre group, six from the polyurethane foam, and six from porcine xenograft group.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
donor sites scar outcome according to a blinded observer | within 9 years after surgery
  evaluated with the scar scale Patient and Observer Scar Assesment Scale (POSAS). The scale contains six items that are scored numerically and when added, constitutes the "Total Score" of the Patient or the Observer Scale. Each of the six items on both scales has a 10-point range (1 - 10), with 10 indicating the worst imaginable scar or sensation. The lowest score, "1" corresponds to the normal skin.
donor sites scar outcome according to a cutometer | within 9 years after surgery
  measurement of elasticity and firmness with cutometer

CONTACTS AND LOCATIONS:
Locations (1):
- The Burn Centre at Linköping University Hospital,, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No